CLINICAL TRIAL: NCT03156530
Title: Auricular Acupuncture Versus Control Group in the Treatment of Balance: a Randomized Controlled Trial
Brief Title: Effect of the Auricular Acupunture of the Lower Limbs on the Equilibrium Response Evaluated by Static Stabilometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tamyris Padovani dos Santos, João Eduardo de Araujo, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 50015413300005440
Record Dates: First submitted 2017-05-05; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2016-03

CONDITIONS: Balance, Postural
Keywords: Acupunture; Acupunture Therapy; Acupunture Points; Acupunture Ear; Postural Balance

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled clinical trial to analyze the influence of auricular points on lower limbs on the equilibrium response assessed by static stabilometry
Masking Description: The subjects were randomized between the groups and the auricular stimulation was performed unilaterally, the motor preference side being standardized as the stimulated side
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auricular acupuncture (Experimental): Stimulated with needles at three joint points of the lower limb, knee and ankle. Balance assessments will be performed prior to (initial) pacing, 20 minutes after the initiation of the pacing protocol (second evaluation) and after 5 minutes the final evaluation.
  Interventions: Device: Auricular acupunture
- Control (Placebo Comparator): Not receive stimulation.
  Interventions: Other: Control

INTERVENTIONS:
Device: Auricular acupunture — Evaluation of balance before, during and after applying of auricular acupuncture.
  Arms: Auricular acupuncture
Other: Control — Not receive stimulation.
  Arms: Control

SUMMARY:
By using a static stabilometry platform, the investigators believe the possible verification of the efficiency of auricular acupuncture points that correlates with regions of our body that may interfere with static equilibrium.

The present work aims to analyze the effect of the stimulation of atrial points of the lower limbs on the equilibrium response evaluated by static stabilometry.

DETAILED DESCRIPTION:
Balance is an extremely relevant subject because of the large and increasing incidence of falls mainly in the elderly population. This leads to a significant social impact since falls can lead an elderly to increasing dependence on the family and can be the cause of depression and reduce their quality of life. Studies have already demonstrated the efficacy of acupuncture stimulation in the treatment of vertigo and also for the improvement of postural control. For this, the option of auricular acupuncture was chosen because it is a non-invasive and safe method. Thus, the objective of this study will be to analyze the effects of atrial stimulation of the lower limbs on the equilibrium response by static stabilometry. Participants in this study were 40 healthy individuals aged between 18 and 30 years who will be divided into two groups: GA (acupuncture group) (n = 20) and CG (control group) (n = 20). The acupuncture group will be stimulated unilaterally according to the motor preference side of each individual in the points referring to the three joints of the lower limb (knee and ankle hip). The control group will not receive stimulation. Balance evaluations will be performed before the stimuation (initial), 20 minutes after the initiation of the protocol (second evaluation) and 5 minutes after the second evaluation, with eyes open and closed. Participants will be positioned standing with their arms along their body, mouth closed not with force and parallel feet. Statistical analysis will be performed by means of a one-way analysis of variance (ANOVA) and the differences between the data will be evidenced by Holm Sidack's post-test. Values of p≤0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 40 healthy individuals between the ages of 18 and 30

Exclusion Criteria:

* Disorders of the central nervous system
* Joint pathologies
* Peripheral neuropathies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of center of force through stabilometry | 1 day
  Evaluation shall be performed during the treatment period.

IPD SHARING:
Plan to Share IPD: No